CLINICAL TRIAL: NCT02398877
Title: Altered Hypothalamic-Pituitary-Adrenal Axis (HPA-Axis) Activity Due To Early Traumatic Stress and Its Relevance for Metabolic Symptoms
Brief Title: HPA Axis Activity Due To Early Traumatic Stress and Metabolic Symptoms
Acronym: Cort-Metab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Head: Clinical Psychology, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: WI 3396/6-1
Record Dates: First submitted 2015-03-09; First posted 2015-03-26 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Childhood Trauma; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Depression with early trauma (Experimental): stress
  Interventions: Other: stress
- Depression without early trauma (Experimental): stress
  Interventions: Other: stress
- Healthy with early trauma (Experimental): stress
  Interventions: Other: stress
- Healthy without early trauma (Experimental): stress
  Interventions: Other: stress

INTERVENTIONS:
Other: stress

SUMMARY:
This study evaluates the association between early trauma, depression and metabolic symptoms.

DETAILED DESCRIPTION:
Early traumatic stress is associated with alterations of the hypothalamic-pituitary-adrenal axis (HPA-axis) indicated by an increased response to stress, a diminished negative feedback and alterations in expression of glucocorticoid receptors. Patients with a history of childhood trauma are more likely to develop metabolic disorders such as diabetes mellitus type 2 or metabolic syndrome.

The investigators will examine participants with and without early life stress and with and without major depression. The investigators assume that traumatized study participants (1) show an increased endocrine stress reaction to psychosocial stress, (2) display an altered sensitivity of GR, and (3) therefore suffer from an adverse cardiovascular risk profile in comparison to not-traumatized participants.

The investigators study will increase current knowledge on possible sequel of early traumatic stress. The results will lead to a more comprehensive understanding of stress-related eating behaviour and its implications.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MDD and/or experience of early trauma

Exclusion Criteria:

* severe illness,
* control group: no diagnosis of MDD and experience of early trauma

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Endocrine response to stress (salivary cortisol) | 2 hours
  salivary cortisol
glucose to oral glucose tolerance test (plasma insulin) | 2 hours
  plasma glucose
insulin to oral glucose tolerance test (plasma insulin) | 2 hours
  plasma insulin
cortisol to corticotropin releasing factor (salivary cortisol) | 3 hours
  salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Katja Wingenfeld, PhD, Principal Investigator — Charite University
Locations (1):
- Charite University, Berlin, Germany